CLINICAL TRIAL: NCT02460094
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study of Intravenously Administered BMS-986168 in Patients With Progressive Supranuclear Palsy
Brief Title: Multiple Ascending Dose Study of Intravenously Administered BMS-986168 (BIIB092) in Patients With Progressive Supranuclear Palsy
Acronym: CN002-003
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CN002-003
Record Dates: First submitted 2015-05-20; First posted 2015-06-02 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Progressive Supranuclear Palsy
MeSH Terms: conditions — Supranuclear Palsy, Progressive | interventions — gosuranemab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Panel 1: BIIB092/ Placebo (Experimental): BIIB092 or matching placebo administered by intravenous (IV) injection, up to a maximum of 3 doses once every four weeks.
  Interventions: Drug: BIIB092; Drug: Placebo
- Panel 2: BIIB092/ Placebo (Experimental): BIIB092 or matching placebo administered by intravenous (IV) injection, up to a maximum of 3 doses once every four weeks.
  Interventions: Drug: BIIB092; Drug: Placebo
- Panel 3: BIIB092/ Placebo (Experimental): BIIB092 or matching placebo administered by intravenous (IV) injection, up to a maximum of 3 doses once every four weeks.
  Interventions: Drug: BIIB092; Drug: Placebo
- Panel 4: BIIB092/ Placebo (Experimental): BIIB092 or matching placebo administered by intravenous (IV) injection, up to a maximum of 3 doses once every four weeks.
  Interventions: Drug: BIIB092; Drug: Placebo

INTERVENTIONS:
Drug: BIIB092 — See Arm Descriptions for dosing information.
  Other Names: BMS-986168
Drug: Placebo — See Arm Descriptions for dosing information. (0.9% Sodium Chloride for Injection or 5% Dextrose Injection if Sodium Chloride is not available)

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of multiple ascending intravenous infusions of BMS-986168 and to assess the pharmacokinetics and immunogenicity of BIIB092, and pharmacodynamics of BIIB092 on cerebrospinal fluid (CSF) extracellular tau (eTau) concentrations in participants with Progressive Supranuclear Palsy.

DETAILED DESCRIPTION:
This study, previously posted by Bristol-Myers Squibb, has transitioned to Biogen under a licensing agreement.

ELIGIBILITY:
Inclusion Criteria

1. Probable or possible PSP defined as:

   * at least a 12-month history of postural instability or falls during the first 3 years that symptoms are present
   * a decreased downward saccade velocity at screening defined as observable eye movement deviation from the "main sequence" linear relationship between saccade amplitude and saccade velocity; or supranuclear ophthalmoplegia defined as 50% reduction in upward gaze or 30% reduction in downward gaze; and
   * age at symptom onset of 40 to 85 years by history and current age between 41 and 86 years, inclusive, at the time of screening; and
   * an akinetic-rigid syndrome with prominent axial rigidity.
   * presence of symptoms for less than 5 years.
2. Body weight range of ≥ 43 kg/95 lbs to ≤ 118 kg/260 lbs.
3. Able to tolerate MRI.
4. Able to perform all protocol-specified assessments and comply with the study visit schedule.
5. Have reliable caregiver to accompany patient to all study visits. Caregiver must be able to read, understand, and speak local language fluently to ensure comprehension of informed consent and informant-based assessments of patient. Caregiver must also have frequent contact with patient (at least 3 hours per week at one time or at different times) and be willing to monitor the patient's health and concomitant medications throughout the study.
6. Score ≥ 20 on the Mini Mental State Exam (MMSE) at screening.
7. Patient must reside outside a skilled nursing facility or dementia care facility at the time of screening, and admission to such a facility is not planned. Residence in an assisted living facility is allowed.
8. Ability to ambulate independently or with assistance defined as the ability to take at least 5 steps with a walker (guarding is allowed provided there is no contact) or the ability to take at least 5 steps without a walker or cane with the assistance of another person who can only have contact with one upper extremity.
9. Stable on other chronic medications for at least 30 days prior to screening.
10. Women of child bearing potential (WOCBP) and sexually active fertile men with partners who are WOCBP must use highly effective birth control.

Exclusion Criteria

1. Presence of other significant neurological or psychiatric disorders.
2. History of or screening brain MRI scan indicative of significant abnormality.
3. History of cancer within 5 years of screening with the exception of fully excised non-melanoma skin cancers or non-metastatic prostate cancer that has been stable for at least 6 months.
4. History of clinically significant hematological, endocrine, cardiovascular, renal, hepatic, gastrointestinal, or neurological disease.
5. Inability to be venipunctured and/or tolerate venous access.
6. Contraindication to undergoing an LP.
7. Recent drug or alcohol abuse as defined in DSM IV.
8. Treatment with any investigational drugs (including placebo) or devices within 90 days prior to screening.
9. Contraindication to the MRI examination for any reason
10. History of a clinically significant medical condition that would interfere with the patient's ability to comply with study instructions, would place the patient at increased risk, or might confound the interpretation of the study results.
11. History of allergy, hypersensitivity, or serious adverse reaction to monoclonal antibodies or related compounds or allergy to any of the components of the study drug

Ages: 41 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-10-02 (Actual); Primary Completion 2016-10-19 (Actual); Study Completion 2016-10-19 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability as Measured by Percentage of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 - Day 169

SECONDARY OUTCOMES:
Percent Change from Baseline in Extracellular Tau (eTau) Concentration in Cerebrospinal Fluid | Day 1 - Day 85
Immunogenicity of BIIB092 Measured by Presence or Absence of Anti-BIIB092 Antibodies in Serum | Day 1 - Day 169
Maximum Serum Concentration (Cmax) of BIIB092 | Day 1 - Day 196
Area Under the Concentration Time-curve of BIIB092 in One Dosing Interval (AUC(TAU)) | Day 1 - Day 196
Trough Serum Concentration (Ctrough) of BIIB092 | Day 1 - Day 196
Serum Concentration at 4 Weeks After Dosing of BIIB092 | Day 1 - Day 196
Time of Maximum Serum Concentration (Tmax) | Day 1 - Day 196

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (13):
- United States (13):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - University of California San Diego, San Diego, California
  - University of California, San Francisco, Medical Center at Parnassus, San Francisco, California
  - Parkinsons Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - University of Florida College of Medicine, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - The University of Chicago Department of Neurology, Chicago, Illinois
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Columbia University Medical Center, New York, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Derived] Boxer AL, Qureshi I, Ahlijanian M, Grundman M, Golbe LI, Litvan I, Honig LS, Tuite P, McFarland NR, O'Suilleabhain P, Xie T, Tirucherai GS, Bechtold C, Bordelon Y, Geldmacher DS, Grossman M, Isaacson S, Zesiewicz T, Olsson T, Muralidharan KK, Graham DL, O'Gorman J, Haeberlein SB, Dam T. Safety of the tau-directed monoclonal antibody BIIB092 in progressive supranuclear palsy: a randomised, placebo-controlled, multiple ascending dose phase 1b trial. Lancet Neurol. 2019 Jun;18(6):549-558. doi: 10.1016/S1474-4422(19)30139-5. PMID 31122495